CLINICAL TRIAL: NCT06507085
Title: Dosimetric Reference Levels for Radioguided Interventional Procedures in Rhythmology. The NR-Rythmo Study
Brief Title: Dosimetric Reference Levels for Radioguided Interventional Procedures in Rhythmology.
Acronym: NR-Rythmo
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2023-2/JG-01
Record Dates: First submitted 2024-07-03; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Radiology, Interventional; Heart Rhythm Disorders
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing radio-guided interventional radiology: All patients undergoing interventional radiology to correct heart rhythm disorders
  Interventions: Radiation: Radio-guided interventions to correct heart rhythm disorders

INTERVENTIONS:
Radiation: Radio-guided interventions to correct heart rhythm disorders — All patients in the cohort will be undergoing one of the following radio-guided procedures :
  * Insertion of a single-chamber pacemaker with lead
  * Insertion of a dual-chamber pacemaker with lead
  * Implantation of a multi-site pacemaker
  * Implantation of a single-chamber endovascular defibrillator
  * Implantation of a dual-chamber endovascular defibrillator
  * Placement of multi-site defibrillator
  * Typical Primary Atrial Flutter Ablation: Cavotricuspid Isthmus only
  * Primo Ablation tachycardia by intra nodal re-entry
  * Accessory pathway ablation
  * Paroxysmal atrial fibrillation ablation (4 pulmonary veins only, all technologies combined
  * Primo Ablation Persistent atrial fibrillation (4 pulmonary veins ± lines ± substrate

SUMMARY:
Interventional radiology has become a widespread technique used in various fields of medicine to diagnose or treat numerous pathologies. However, the risk of X-rays must be taken into account. In 2019, the French Authority on Nuclear Safety published diagnostic reference levels for radio-guided interventional practices for 10 interventional radiology procedures and 2 interventional cardiology procedures, based on studies published by the French Society of Medical Physics in collaboration with the French Society of Radiology and the French Coronary Artery Disease and Interventional Cardiology Group. Reference levels for interventional procedures under CT guidance were also defined in 2020 following a national multicenter study coordinated by Nîmes University Hospital (NIMAO NRD-SI). However, no national multicentre studies have ever defined reference levels for radioguided interventional procedures in rhythmology. The aim of this study is to define standard national dosimetric levels for a number of radioguided interventional procedures in rhythmology.

DETAILED DESCRIPTION:
Interventional radiology has become a widespread technique used in various fields of medicine to diagnose or treat numerous pathologies. However, the risk of X-rays must be taken into account.

To provide healthcare professionals with an optimization tool, the International Commission on Radiological Protection (ICRP) introduced the concept of diagnostic reference levels (DRLs) in 1997. For the first time, in 2019, the French Authority on Nuclear Safety published DRLs for radio-guided interventional practices for 10 interventional radiology procedures and 2 interventional cardiology procedures, based on studies published by the French Society of Medical Physics in collaboration with the French Society of Radiology and the French Coronary Artery Disease and Interventional Cardiology Group. Reference levels for interventional procedudures under CT guidance were also defined in 2020 following a national multicentre study coordinated by Nîmes University Hospital (NIMAO NRD-SI). However, no national multicentre studies have ever defined reference levels for radioguided interventional procedures in rhythmology. The aim of this study is to define standard national diagnostic reference levels for radioguided interventional procedures in rhythmology for the following acts:

* Insertion of a single-chamber pacemaker with lead (DELF 007 according to the common French classification for medical acts)
* Insertion of a dual-chamber pacemaker with lead (DELF 005 according to the common French classification for medical acts)
* Implantation of a multi-site pacemaker (DELF 001 and/or DELF 015 according to the common French classification for medical acts)
* Implantation of a single-chamber endovascular defibrillator (DELF 013 according to the common French classification for medical acts)
* Implantation of a dual-chamber endovascular defibrillator (DELF 015 according to the common French classification for medical acts)
* Placement of multi-site defibrillator (DELF 020 or DELF 014 according to the common French classification for medical acts)
* Typical Primary Atrial Flutter Ablation: Cavotricuspid Isthmus only (DEPF 012 according to the common French classification for medical acts)
* Primo Ablation tachycardia by intra nodal re-entry (DEPF 010 according to the common French classification for medical acts)
* Accessory pathway ablation (DEPF 005 according to the common French classification for medical acts)
* Paroxysmal atrial fibrillation ablation (4 pulmonary veins only, all technologies combined; DEPF 033 as per the common French classification for medical acts)
* Primo Ablation Persistent atrial fibrillation (4 pulmonary veins ± lines ± substrate; DEPF 033 ± DEPF 014 ± DENF 018 ± DEPF 012 according to the common French classification for medical acts) Secondaires objectives include the evaluation of interventional practices for each procedure performed regarding the use of a fixed or mobile C-arm, the make, model and year of installation of the equipment used, deviation at last external quality control between displayed and measured dose area product and, if available, between displayed and measured Kair, the lowest/highest scan rates used during the procedure, use of graphy,lowest/highest scan rate(s) used during procedures, use of collimation during procedures, use of a 3D mapping system, the type of technique used for an ablation procedure, if used, the use of a cage-type radiation protection system during the procedure, cone beam computed tomography performed during procedure, CT scan before the procedure, duration of the procedure and the experience of the operator performing the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Adult male/female patient (≥ 18 years)
* Body Mass Index (BMI) between 18 and 35 kg/m².
* Patient to benefit from one of the following procedures:

Placement of single-chamber pacemaker with lead (DELF 007 according to CCAM) Dual-chamber pacemaker insertion with lead (DELF 005 according to CCAM) Multi-site pacemaker placement (DELF 001 and/or DELF 015 according to CCAM) Placement of single-chamber endovascular defibrillator (DELF 013 according to CCAM) Placement of dual-chamber endovascular defibrillator (DELF 015 according to CCAM) Placement of multi-site defibrillator (DELF 020 or DELF 014 according to CCAM) Primo Ablation Typical Atrial Flutter: Cavotricuspid Isthmus only (DEPF 012 according to CCAM) Primo Ablation tachycardia by intra nodal re-entry (DEPF 010 according to CCAM) Accessory pathway ablation (DEPF 005 according to CCAM) Paroxysmal atrial fibrillation ablation (4 pulmonary veins only, all technologies combined; DEPF 033 as per CCAM) Primo Ablation Persistent atrial fibrillation (4 pulmonary veins ± lines ± substrate; DEPF 033 ± DEPF 014 ± DENF 018 ± DEPF 012 according to CCAM)

Exclusion Criteria:

* Patient whose procedure does not require X-rays
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population: All patients benefitting from a rhythmology procedure to be performed among the procedures defined in the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 6600 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Radiation dose: Insertion of a single-chamber pacemaker with lead (DELF 007 according to the common French classification for medical procedures) | Day 1 of the intervention
  Total Dose Area Product for the procedure measured in Gy.cm2
Total Air Kerma: Insertion of a single-chamber pacemaker with lead (DELF 007 according to the common French classification for medical procedures) | Day 1 of the intervention
  The total Air Kerma for the procedure will be measured at the interventional reference point (Kair) in Gy
Total scanning time: Insertion of a single-chamber pacemaker with lead (DELF 007 according to the common French classification for medical procedures) | Day 1 of the intervention
  The total scanning time for the procedure will be measured in seconds
Total number of images: Insertion of a single-chamber pacemaker with lead (DELF 007 according to the common French classification for medical procedures) | Day 1 of the intervention
  Quantitative
Radiation dose: Insertion of a dual-chamber pacemaker with lead (DELF 005 according to the common French classification for medical acts | Day 1 of the intervention
  Total Dose Area Product for the procedure measured in Gy.cm2
Total Air Kerma: Insertion of a dual-chamber pacemaker with lead (DELF 005 according to the common French classification for medical acts | Day 1 of the intervention
  The total Air Kerma for the procedure will be measured at the interventional reference point (Kair) in Gy
Total scanning time: Insertion of a dual-chamber pacemaker with lead (DELF 005 according to the common French classification for medical acts | Day 1 of the intervention
  The total scanning time for the procedure will be measured in seconds
Total number of images: Insertion of a dual-chamber pacemaker with lead (DELF 005 according to the common French classification for medical acts | Day 1 of the intervention
  Quantitative
Radiation dose: Implantation of a multi-site pacemaker (DELF 001 and/or DELF 015 according to the common French classification for medical acts) | Day 1 of the intervention
  Total Dose Area Product for the procedure measured in Gy.cm2
Total Air Kerma: Implantation of a multi-site pacemaker (DELF 001 and/or DELF 015 according to the common French classification for medical acts) | Day 1 of the intervention
  The total Air Kerma for the procedure will be measured at the interventional reference point (Kair) in Gy
Total scanning time: Implantation of a multi-site pacemaker (DELF 001 and/or DELF 015 according to the common French classification for medical acts) | Day 1 of the intervention
  The total scanning time for the procedure will be measured in seconds
Total number of images: Implantation of a multi-site pacemaker (DELF 001 and/or DELF 015 according to the common French classification for medical acts) | Day 1 of the intervention
  Quantitative
Radiation dose: Implantation of a single-chamber endovascular defibrillator (DELF 013 according to the common French classification for medical acts) | Day 1 of the intervention
  Total Dose Area Product for the procedure measured in Gy.cm2
Total Air Kerma: Implantation of a single-chamber endovascular defibrillator (DELF 013 according to the common French classification for medical acts) | Day 1 of the intervention
  The total Air Kerma for the procedure will be measured at the interventional reference point (Kair) in Gy
Total scanning time: Implantation of a single-chamber endovascular defibrillator (DELF 013 according to the common French classification for medical acts) | Day 1 of the intervention
  The total scanning time for the procedure will be measured in seconds
Total number of images: Implantation of a single-chamber endovascular defibrillator (DELF 013 according to the common French classification for medical acts) | Day 1 of the intervention
  Quantitative
Radiation dose: Implantation of a dual-chamber endovascular defibrillator (DELF 015 according to the common French classification for medical acts) | Day 1 of the intervention
  Total Dose Area Product for the procedure measured in Gy.cm2
Total Air Kerma: Implantation of a dual-chamber endovascular defibrillator (DELF 015 according to the common classification for medical acts) | Day 1 of the intervention
  The total Air Kerma for the procedure will be measured at the interventional reference point (Kair) in Gy
Total scanning time: Implantation of a dual-chamber endovascular defibrillator (DELF 015 according to the common French classification for medical acts) | Day 1 of the intervention
  The total scanning time for the procedure will be measured in seconds
Total number of images: Implantation of a dual-chamber endovascular defibrillator (DELF 015 according to the common French classification for medical acts) | Day 1 of the intervention
  Quantitative
Radiation dose: Placement of multi-site defibrillator (DELF 020 or DELF 014 according to the common French classification for medical acts) | Day 1 of the intervention
  Total Dose Area Product for the procedure measured in Gy.cm2
Total Air Kerma : Placement of multi-site defibrillator (DELF 020 or DELF 014 according to the common French classification for medical acts) | Day 1 of the intervention
  The total Air Kerma for the procedure will be measured at the interventional reference point (Kair) in Gy
Total scanning time: Placement of multi-site defibrillator (DELF 020 or DELF 014 according to the common French classification for medical acts) | Day 1 of the intervention
  The total scanning time for the procedure will be measured in seconds
Total number of images: Placement of multi-site defibrillator (DELF 020 or DELF 014 according to the common French classification for medical acts) | Day 1 of the intervention
  Quantitative
Radiation dose : Primary Atrial Flutter Ablation: Cavotricuspid Isthmus only (DEPF 012 according to the common French classification for medical acts) | Day 1 day of the intervention
  Total Dose Area Product for the procedure measured in Gy.cm2
Total Air Kerma: Primary Atrial Flutter Ablation: Cavotricuspid Isthmus only (DEPF 012 according to the common French classification for medical acts) | Day 1 of the intervention
  The total Air Kerma for the procedure will be measured at the interventional reference point (Kair) in Gy
Total scanning time: Primary Atrial Flutter Ablation: Cavotricuspid Isthmus only (DEPF 012 according to the common French classification for medical acts) | Day 1 of the intervention
  The total scanning time for the procedure will be measured in seconds
Total number of images: Primary Atrial Flutter Ablation: Cavotricuspid Isthmus only (DEPF 012 according to the common French classification for medical acts) | Day 1 of the intervention
  Quantitative
Radiation dose: Primo Ablation tachycardia by intra nodal re-entry (DEPF 010 according to the common French classification for medical acts) | Day 1 of the intervention
  Total Dose Area Product for the procedure measured in Gy.cm2
Total Air Kerma: Primo Ablation tachycardia by intra nodal re-entry (DEPF 010 according to the common French classification for medical acts) | Day 1 of the intervention
  The total Air Kerma for the procedure will be measured at the interventional reference point (Kair) in Gy
Total scanning time: Primo Ablation tachycardia by intra nodal re-entry (DEPF 010 according to the common French classification for medical acts) | Day 1 of the intervention
  The total scanning time for the procedure will be measured in seconds
Total number of images: Primo Ablation tachycardia by intra nodal re-entry (DEPF 010 according to the common French classification for medical acts) | Day 1 of the intervention
  Quantitative
Radiation dose: pathway ablation (DEPF 005 according to the common French classification for medical acts) | Day 1 of the intervention
  Total Dose Area Product for the procedure measured in Gy.cm2
Total Air Kerma: pathway ablation (DEPF 005 according to the common French classification for medical acts) | Day 1 of the intervention
  The total Air Kerma for the procedure will be measured at the interventional reference point (Kair) in Gy
Total scanning time: pathway ablation (DEPF 005 according to the common French classification for medical acts) | Day 1 of the intervention
  The total scanning time for the procedure will be measured in seconds
Total number of images: pathway ablation (DEPF 005 according to the common French classification for medical acts) | Day 1 of the intervention
  Quantitative
Radiation dose: Paroxysmal atrial fibrillation ablation (4 pulmonary veins only, all technologies combined; DEPF 033 as per the common French classification for medical acts) | Day 1 of the intervention
  Total Dose Area Product for the procedure measured in Gy.cm2
Total Air Kerma: Paroxysmal atrial fibrillation ablation (4 pulmonary veins only, all technologies combined; DEPF 033 as per the common French classification for medical acts) | Day 1 of the intervention
  The total Air Kerma for the procedure will be measured at the interventional reference point (Kair) in Gy
Total scanning time: Paroxysmal atrial fibrillation ablation (4 pulmonary veins only, all technologies combined; DEPF 033 as per the common French classification for medical acts) | Day 1 of the intervention
  The total scanning time for the procedure will be measured in seconds
Total number of images: Paroxysmal atrial fibrillation ablation (4 pulmonary veins only, all technologies combined; DEPF 033 as per the common French classification for medical acts) | Day 1 of the intervention
  Quantitative
Radiation dose: Primo Ablation Persistent atrial fibrillation (4 pulmonary veins ± lines ± substrate; DEPF 033 ± DEPF 014 ± DENF 018 ± DEPF 012 according to the common French classification for medical acts) | Day 1 of the intervention
  Total Dose Area Product for the procedure measured in Gy.cm2
Total Air Kerma: Primo Ablation Persistent atrial fibrillation (4 pulmonary veins ± lines ± substrate; DEPF 033 ± DEPF 014 ± DENF 018 ± DEPF 012 according to the common French classification for medical acts) | Day 1 of the intervention
  The total Air Kerma for the procedure will be measured at the interventional reference point (Kair) in Gy
Total scanning time: Primo Ablation Persistent atrial fibrillation (4 pulmonary veins ± lines ± substrate; DEPF 033 ± DEPF 014 ± DENF 018 ± DEPF 012 according to the common French classification for medical acts) | Day 1 of the intervention
  The total scanning time for the procedure will be measured in seconds
Total number of images: Primo Ablation Persistent atrial fibrillation (4 pulmonary veins ± lines ± substrate; DEPF 033 ± DEPF 014 ± DENF 018 ± DEPF 012 according to the common French classification for medical acts) | Day 1 of the intervention
  Quantitative

SECONDARY OUTCOMES:
Use of a fixed or mobile C-arm in each of the above 11 interventions | Day 1 of the intervention
  YES /NO
Equipment | Day 1 of the intervention
  The make, model and year of commissioning the C-arm used will be recorded.
Deviation between the Dose Area Product displayed and measured | Day 1 of the intervention
  The date of the last mandatory Quality Control and deviation between the Dose Area Product displayed and actually measured will be recorded.
Deviation between the total air Kerma displayed and measured | Day 1 of the intervention
  The date of the last mandatory Quality Control and deviation between the total air Kerma displayed and actually measured will be recorded.
Lowest/highest fluoroscopy frame rates | Day 1 of the intervention
  The lowest/highest frame rates used during fluoroscopy procedures will be measured in p/s
Use of fluorography | Day 1 of the intervention
  YES/NO
Lowest /highest fluorography rates | Day 1 of the intervention
  The lowest/highest frame rates used during fluorography procedures will be measured in p/s
Use of collimation during each of the above 11 procedures ? | Day 1 of the intervention
  YES/NO
Use of a 3D mapping system during each of the above 11 procedures ? | Day 1 of the intervention
  YES/NO
Technique used for ablation | Day 1 of the intervention
  The type of technique used for ablation procedures will be recorded
Use of a collective radiation protection system during each of the above 11 procedures ? | Day 1 of the intervention
  YES/NO
Cone Beam Computed Tomography performed during any of the procedures above ? | Day 1 of the intervention
  YES/NO
CT scan before a paroxysmal atrial fibrillation ablation procedure ? | Day 1 of the intervention
  YES/NO
Duration of each of the above procedures | Day 1 of the intervention
  The duration of each of the above procedures will be recorded in minutes
Rhythmologist's experience | Day 1 of the intervention
  The number of years of experience of the surgeon who performed the procedure will be recorded in years

CONTACTS AND LOCATIONS:
Overall Officials: Pierre François Winum, Dr., Principal Investigator — Nîmes University Hospital
Locations (1):
- Nîmes University Hospital, Nîmes, Gard, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Amara W, Socie P, Renault C, Taieb J. [Where are done electrophysiology procedures in France and what is the expected evolution ?]. Ann Cardiol Angeiol (Paris). 2022 Nov;71(5):294-298. doi: 10.1016/j.ancard.2022.08.010. French. PMID 36424019
- [Background] Etard C, Bigand E, Salvat C, Vidal V, Beregi JP, Hornbeck A, Greffier J. Patient dose in interventional radiology: a multicentre study of the most frequent procedures in France. Eur Radiol. 2017 Oct;27(10):4281-4290. doi: 10.1007/s00330-017-4780-5. Epub 2017 Mar 13. PMID 28289939
- [Background] Greffier J, Ferretti G, Rousseau J, Andreani O, Alonso E, Rauch A, Gillet R, Le Roy J, Cabrol-Faivre L, Douane F, David A, Henry S, Jacques T, Stefanovic X, Decoux E, Lafay F, Pilleul F, Couzon F, Boutet C, Woerly B, Baur P, Sans N, Faruch M, Moussier-Lherm A, Tselikas L, Jacquier A, Bigand E, Pessis E, Teriitehau C, Magnier F, Cassagnes L, Haberlay M, Boutteau D, De Kerviler E, Majorel-Gouthain C, Defez D, Vuillod A, Rouviere O, Hennequin L, Fohlen A, Alwan R, Malakhia A, Aubry S, Dohan A, Eresue-Bony M, Gautier R, Dal R, Dabli D, Hebert T, Kovacs R, Hadid-Beurrier L, Bousson V, Potel M, Barbotteau Y, Michel C, Habib-Geryes B, Andre M, Arnaud T, Bestion N, Ernst O, Monfraix S, Brillet PY, Guiu B, Boussel L, Demonchy M, Beregi JP, Frandon J. National dose reference levels in computed tomography-guided interventional procedures-a proposal. Eur Radiol. 2020 Oct;30(10):5690-5701. doi: 10.1007/s00330-020-06903-9. Epub 2020 May 2. PMID 32361774
- [Background] Bar O, Maccia C, Pages P, Blanchard D. A multicentre survey of patient exposure to ionising radiation during interventional cardiology procedures in France. EuroIntervention. 2008 Mar;3(5):593-9. doi: 10.4244/eijv3i5a107. PMID 19608487
- [Background] Radiological protection and safety in medicine. A report of the International Commission on Radiological Protection. Ann ICRP. 1996;26(2):1-47. No abstract available. PMID 8911634
- [Background] Diagnostic reference levels in medical imaging: review and additional advice. Ann ICRP. 2001;31(4):33-52. PMID 12685758